CLINICAL TRIAL: NCT06576609
Title: Effectiveness of INJEX Versus Traditional Syringe During Restoration of Primary Teeth: A Randomized Split-mouth Clinical Trial
Brief Title: Effectiveness of INJEX Versus Traditional Syringe During Restoration of Primary Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jazan (Other Government)
Responsible Party: Principal Investigator, satish vishwanathaiah, Associate Professor, University of Jazan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: University Jazan
Record Dates: First submitted 2024-08-26; First posted 2024-08-29 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Child Behavior
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INJEX (Experimental): Needle less device
  Interventions: Device: INJEX [ Needle less anesthesia]
- Needle syringe (Active Comparator): traditional dental needle
  Interventions: Device: INJEX [ Needle less anesthesia]

INTERVENTIONS:
Device: INJEX [ Needle less anesthesia] — already described
  Other Names: Syringe Needle [ Traditional technique]

SUMMARY:
The main purpose of this study is to make a comparison between pain perception levels and the behavior of patients during the restoration process in children between a needleless local anesthetic system (INJEX) and the conventional syringe technique. The main purpose of this study is to make a comparison between pain perception levels and the behavior of patients during the restoration process in children between a needleless local anesthetic system (INJEX) and the conventional syringe technique.

. The main questions it aims to answer are:

1. To evaluate pain perception for restoration of primary molars with a needle free system in a pediatric population.
2. To evaluate pain perception for restoration of Primary molars with needle syringe [Traditional syringe system] method in a pediatric population
3. Time required to deliver anesthesia using needle free system vs Needle syringe [ traditional syringe system] Participants who enrolled in the study will be anesthetized according to the respective groups i,e INJEX (needle free system) and traditional dental needle system and restoration will be done.

DETAILED DESCRIPTION:
Before the start of the study a written informed consent and ascent was obtained from each parent of the children included in the study stating they accepted the treatment. Ethical clearance will be obtained before the start of the study. Patients reporting to the dental clinics, college of dentistry will be included in the study.

Sample size estimation:

The sample size was determined using the following formula, based on a difference in mean Face, Legs, Activity, Cry, and Consolability (FLACC) scores of 1.2 and a pooled standard deviation of 1.89. Sample Size (n) = 2Sp2 (Z 1-α/2+Z1-β) 2 µd2 where, Z (1-α/2) = 1.96 for a 95% confidence interval Z1-β = 0.84 for 80% power Sp2 = pooled standard deviation µd = 1.2 (difference in mean between groups) Substituting these values, the sample size was estimated to be 21. An additional 20% of the estimated sample size was added to account for any potential sampling loss, bringing the final sample size to a total of 25 teeth in each group.

study design: It was a split mouth randomized controlled trial

Randomization:

Teeth designated for restoration were assigned to one of two groups using a simple randomization method with a 1:1 allocation ratio. The allocation was performed using a predetermined list, with the first list for the right side, and the second for the left side. Allocation concealment was maintained through sealed envelopes until the time of intervention to prevent selection bias. On the intervention day, patients identified their number on either the right or left side lists.

Group I: All teeth in this group underwent restoration using the traditional syringe system. Making use of a conventional syringe fitted with a 27-gauge needle (Hogen Spitze, C-K Dental IND.CO., LTD.) local infiltration of Scandicaine 2% Special (mepivacaine hydrochloride and adrenaline) was given.

Group II: Teeth in this group received treatment with the needle-free injection system, INJEX (INJEX Pharma AG, Germany).

Intervention procedure To mitigate any operator-related bias, a single operator conducted the entire anesthesia protocol for all participants in the trial. Utilizing the "Tell-Show-Do" technique, all relevant treatment equipment and protocols were introduced and explained. The injection was thoroughly described using appropriate euphemisms or age-appropriate language.

A sterile dry gauze was used to cleanse the treatment area at the injection site before administering LA. Following this, a very small quantity of topical anesthetic (Benzocaine 20%, NJ, USA) was given and left to remain for a minimum time of 1 minute. Following the application of topical anesthesia, LA was administered based on the participant's assigned group.

After a standard waiting time of 3 minutes for the anesthesia to take effect, dental caries were removed , The pulp capping material, Dycal (Dentsply Caulk, Milford, DE, USA), was placed, and a type IX glass ionomer cement (GC Corporation, Tokyo, Japan) liner was applied before the final restoration with composite material.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 7 - 10 years
* Existence of deep carious Primary molar, indicated for Indirect pup capping.
* Complete physical and mental health without any confounding medical history
* Parents who gave written informed consent

Exclusion Criteria:

* Children below 7 years of age
* Children complaining of irreversible pulpitis.
* Children with Negative behaviour according to the wright's modification of
* Frankl Behaviour Rating scale (FBRS) during initial examination
* Children with medical or mentally compromised

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2024-02-16 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
The Face, Legs, Activity, Cry, and Consolability (FLACC) Scale | during and immediately after the delivery of anesthesia
  FLACC gives an observational pain scale during the delivery of anesthesia

SECONDARY OUTCOMES:
Frankel Behaviour Rating Scale ( FBRS) | before the delivery of anesthesia, during the delivery of anesthesia and after the delivery of anesthesia
  Frankel 1 -- definitely negative, Frankel 2 - Negative, Frankel 3 - positive, Frankel 4 - Definitely positive
Pulse rate | Before the delivery of anesthesia, immediately after the delivery of anesthesia, and 1 minute after the delivery of anesthesia
  comfort and patient acceptance during treatment
Wong Baker Scale | During and immediately after the delivery of anesthesia
  Used to self-assess and effectively communicate the severity of pain they may be experiencing
Time of local anesthesia administration | during the delivery of anesthesia
  comfort and patient acceptance during treatment

CONTACTS AND LOCATIONS:
Locations (1):
- College of Dentistry, Jizan, Jazan Region, Saudi Arabia